CLINICAL TRIAL: NCT03656276
Title: The "ToPIC" Study = Tool to Improve Participation In Clinical Trials
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: UW16060; 2016-1579 (Other: Health Science Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); P30CA014520 (NIH)
Record Dates: First submitted 2018-08-28; First posted 2018-09-04 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Communication; Physician-Patient Relations
MeSH Terms: conditions — Communication | interventions — Clinical Trials as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Oncologists (wait list control): Oncologists will be wait-listed for training on the Tool to improve Participation In Clinical Trials (ToPIC)
- Group B: Oncologists (training): Oncologists will receive immediate training on the Tool to improve Participation In Clinical Trials (ToPIC)
  Interventions: Behavioral: Tool to improve Participation In Clinical Trials (ToPIC)

INTERVENTIONS:
Behavioral: Tool to improve Participation In Clinical Trials (ToPIC) — The Tool to improve Participation In Clinical Trials (ToPIC) is a communication tool to facilitate clinical trial decision making conversations between oncologists and patients.
  Groups: Group B: Oncologists (training)

SUMMARY:
The purpose of this study is to pilot the "ToPIC" tool, a communication tool to facilitate clinical trial decision making conversations between oncologists and patients.

DETAILED DESCRIPTION:
The ToPIC tool is a structured delivery of important treatment-related information. The oncologist remains entirely in charge of the information delivered (e.g. what are the treatment options, what are the potential benefits) and uses the ToPIC framework to organize the information and create a pen and paper diagram for the patient to assist in their processing and deliberation. The tool creates a forum for a clear presentation of options and facilitates a patient's ability to express their individual preferences.

Oncologists are the intervention population and will be trained in how to use the ToPIC communication tool. Volunteer oncologists will be randomly assigned to immediate training or wait list control. Oncologists who are randomly assigned to the intervention group will receive training, and once they have demonstrated competence with the tool, they will begin using the tool with their patients. Data collection for any patient whom they present treatment options which include a clinical trial will be included for the primary analysis related to recruitment for clinical trials. This collection will begin once the oncologist, regardless of their assigned group, has signed consent and been randomized.

ELIGIBILITY:
Inclusion Criteria:

* (Oncologists) - All UW Health oncologists who engage with patients about treatment decisions which involve therapeutic clinical trials. Eligible oncologists may work at UW Hospital and 1 South Park and include all medical, radiation and surgical oncologists. Participation by oncologists is completely voluntary.
* (Patients)

  * Any adults (over age 18)
  * Seen in any UW oncology clinic
  * Participated in a discussion with a participating oncologist about treatment options that included a therapeutic clinical trial.

Exclusion Criteria:

* (Oncologists) ToPIC Study PI
* (Patients) Non-English speaking patients. We exclude non-english speakers due to the unpredictable impacts of the translation/interpreter dynamic and the lack of a pen/paper diagram in the patient's native language. This would include deaf patients.

  * Blind patients (or someone who cannot see the pen/paper diagram)
  * Those who do not have capacity for decision making.
  * Those offered participation in non-therapeutic intent clinical trials. This would include Phase 1 clinical trials due to the non-therapeutic intent.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: UW Health Oncologists and their Patients
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients that consent to a therapeutic trial. | may be up to 4 months following appointment with Oncologist
  Number of patients that consent to a therapeutic trial in the wait-list control vs. the trained oncologist groups. Per protocol, there is no timeframe within which patients need to consent. Due to the nature of oncology care, some patients are presented with the trial months before they are eligible, and the team follows up to see if they choose to consent if/when they are eligible.

SECONDARY OUTCOMES:
Number of oncologists that can learn the ToPIC tool after 3 hours of training. | At completion of 3-hour training
  Oncologists will demonstrate their post-training competence with a standardized patient-actor encounter. Competency is assessed by a 4-person panel using a 20-point scoring system. A consensus score of 14 or above indicates competency.
Number of patients that enroll in a therapeutic trial. | may be up to 6 months following consent
  Number of patients that enroll in a therapeutic trial in the wait-list control vs. the trained oncologist groups. Per protocol, there is no timeframe within which patients need to enroll. Enrollment in the trial may be prolonged due to extensive screening requirements.
Number of patients that agree to hear about therapeutic trial. | up to 18 months
  Number of patients that agree to hear about therapeutic trial in the wait-list control vs. the trained oncologist groups. Physicians will be on study for up to 18 months once they are trained (ToPIC trained group) or enrolled (waitlist control group). The number of patients who agree to hear about the trial will be collected during the 18 month period.

OTHER OUTCOMES:
Qualitative interviews with patients and clinicians to assess the acceptability of ToPIC conversation. | Within 12 weeks following oncology appointment.
  Interviews to better understand the factors that clinicians and patients consider when making treatment decisions about clinical trials and their impression of the decision making discussion.

CONTACTS AND LOCATIONS:
Overall Officials: Toby Campbell, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/